CLINICAL TRIAL: NCT06102304
Title: Effect of Focused Focused Extracorpeal Shock Wave on the Myo-Electrical and Nerve Root Function in Patients With Cervical Radiculopathy
Brief Title: Myo-Electrical and Nerve Root Function Response to Focused Extracorpeal Shock Wave in Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Badreldin Saleh Moustafa, PhD, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004747
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-11

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy; Nerve root Dysfunction; Trigger points; Focused Extracorpeal Shock Wave
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical trial, where the recruited patients will be randomly assigned into 2 equal groups ( GA & GB) using sealed envelopes. Control group (GA) and study group (GB). Patients in (GA) will be treated by a designed physiotherapy program consisted of Myo-facial release, stretching exercise, Proprioceptive neuromuscular facilitation (PNF) techniques, Median nerve glide techniques ,Graduated strengthening exercises for the upper limb, exercises in addition to sham shock wave on the upper trapezius. Patients in (GB) will be treated by focused Extracorpeal shock wave on the trigger points of upper trapezius in addition to the same physiotherapy program as GA.
Who Masked: Participant
Masking Description: Patients participated will be masked about the type of intervention, where (GA) patients will receive PT program + sham shock wave on upper trapezius, while patients in (GB) will receive focused extracorpeal shock wave on the trigger points of upper trapezius in addition to the same PT program as (GA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Extracorpeal Shock Wave (Placebo Comparator): Control group (GA) Patients in (GA) will be treated by a designed physiotherapy program consisted of Myo-fascial release, stretching exercise, Proprioceptive neuromuscular facilitation (PNF) techniques, Median nerve neural glide techniques, Graduated strengthening exercises for the upper limb in addition to sham shockwave on the upper trapezius.
  Interventions: Device: Sham Extracorpeal shock wave
- Focused Extracorpeal Shock wave (Experimental): Patients in (GB) will be treated by Focused Extracorpeal shockwave on the trigger points of upper trapezius in addition to the same physiotherapy program as GA.
  Interventions: Device: Focused Extracorpeal Shock wave

INTERVENTIONS:
Device: Focused Extracorpeal Shock wave — Focused Extracorporeal shock wave for 700 impulses of 0.056 mJ/mm at a frequency of 10 Hz to the taut band and 300 impulses surrounding the taut band was applied as low energy 2 sessions per week for 4 weeks. (EME S.r.l. via Degli Abeti 88/161122 Pesaro [serial number: EM12681015], Italy) was used as a focused extracorporeal shock wave therapy apparatus.
  Arms: Focused Extracorpeal Shock wave
Device: Sham Extracorpeal shock wave — (EME S.r.l. via Degli Abeti 88/161122 Pesaro [serial number: EM12681015], Italy) was used as a focused extracorporeal shock wave therapy apparatus. The device will be used in the demo mood with no radiation or impulses applied.
  Arms: Sham Extracorpeal Shock Wave

SUMMARY:
BACKGROUND: Upper limb nerve root dysfunction with increased active myofascial trigger point in upper trapezius is common problem in patients with cervical radiculopathy.

The purpose of this study was to evaluate the effect of Extracorpeal shock wave on the myo-electric and nerve function responses in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
Randomized controlled clinical trial among Forty eight (48) patients with cervical radiculopathy.

They will be allocated randomly by sealed envelopes into two groups: Group (A): will receive a designed physical therapy program in addition to sham Extracorpeal shock wave on upper trapezius. Group (B): will receive Focused Extracorpeal shock wave on the active myofascial trigger points in upper trapezius in addition to the same physical therapy program as in group A.

Somatosensory evoked potential for upper limb median nerve will be applied using the Electromyography (EMG) device. Hand grip strength will be assessed using the handheld dynamometer (HHD) , Level of radiating pain will be assessed using the numeric rating scale , Pain and tenderness in upper trapezius muscle will be also assessed using Pressure pain threshold (PPT).

ELIGIBILITY:
Inclusion Criteria:

1. All patients suffer from unilateral discogenic cervical radiculopathy of lower cervical spine(C5-C6 and/ or C6-C7) as confirmed with MRI.
2. All patients suffer from pain and tenderness on active trigger points of the upper trapezius .
3. Age ranging from 36 to 46 years old.
4. Duration of symptoms more than 3 months to avoid acute stage of inflammation.
5. Side to side amplitude differences of 50% or more in DSSEPs measurement (Naguszewski et al.,2001)

Exclusion Criteria:

1. Posterior osteophytes
2. Spinal canal stenosis
3. Rheumatoid arthritis
4. Vestibular insufficiency
5. Osteoporosis
6. Any signs or symptoms of myelopathy
7. Any abnormalities of deep sensation
8. Associated pathologies of upper cervical region or the upper limb that may cause overlapping with clinical findings as referred pain from costotransverse joint, rotator cuff tendonitis, cervical rib syndrome and entrapment neuropathy.

Ages: 36 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Amplitude of median nerve dermatomal somatosensory evoked potential | Baseline Assessment and Immediately Post Treatment.
  After the stimulation was performed and the traces were superimposed to ensure reproducibility, negative near field potential were detected and positive peak was detected to measure the peak to peak amplitude. This amplitude was measured. The distance between positive and negative peak , it is measures in millivolts (mV)
Distal Latency of median nerve dermatomal somatosensory evoked potential | Baseline Assessment and Immediately Post Treatment.
  Distal latency is defined as the interval between the stimulation of a compound muscle or selective dermatome and the observed response. It is measured in meter per second (m/s)
Pain Pressure Threshold on upper trapezius | Baseline Assessment and Immediately Post Treatment.
  Pain pressure Threshold (PPT) device will be used to detect tenderness and pain on the active myofascial trigger points on upper trapezius muscle. The 1-cm² rubber tip was applied perpendicularly over the myofascial trigger points and the power is switched on; a required pressure will be exerted on the site of myofascial trigger points by pressing the transducers firmly downwards. Measurements were recorded in kilograms of pressure per square centimeter (kg/cm^2).
Hand grip Strength | Baseline Assessment and Immediately Post Treatment.
  Jamar hydraulic hand dynamometer will be used, it is a quantitative and an objective measure of the isometric muscular strength of the hand grip. It is a portable dynamometer used as a valid and reliable tool to reflect the upper limb strength. This instrument is scored using force production in kilograms (0-90) or pounds (0-200). Maximum grip was the mean of three trials. For each patient the both sides were assessed before treatment to collect the normative value for each patient. Mean of Maximum grip was compared pre and post treatment for each patient
Level of radiating pain | Baseline Assessment and Immediately Post Treatment.
  Numeric rating Scale (NRS) for pain will be used to assess level of pain radiating through the upper limb. Patients are asked to circle the number between 0 and 10 that fits best to their pain intensity . Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.

CONTACTS AND LOCATIONS:
Overall Officials: Engy BadrEldin S Moustafa, PhD, Principal Investigator — Faculty of Physical Therapy, Cairo University, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No